CLINICAL TRIAL: NCT03529214
Title: A Program Evaluation to Measure the Feasibility of the Team Birth Project
Brief Title: An Evaluation of the Team Birth Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Neel Shah, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB18-0550
Record Dates: First submitted 2018-04-16; First posted 2018-05-18 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Complications; Cesarean Section Complications; Maternal Complication of Pregnancy; Communication, Multidisciplinary
Keywords: Quality Improvement; Program Evaluation; Quality Assurance; Feasibility; Acceptability
MeSH Terms: conditions — Pregnancy Complications; Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implemented Health Facility (Other): Health facility that has piloted the "Team Birth Project"
  Interventions: Behavioral: Exposed study site

INTERVENTIONS:
Behavioral: Exposed study site — The study sites will pilot the Team Birth Project designed to improve team communication (between providers, as well as providers and patients). The project includes three key implementation steps that involve: preparing local sites for the implementation of the project; training and coaching on the use of the tools; and sustainment through peer coaching and data feedback. A mixed methods approach will be used to assess acceptability and feasibility, including: (1) clinician surveys and interviews, (2) implementation team focus groups, and (3) patient surveys.

SUMMARY:
The purpose of this study is to evaluate the feasibility of a pilot project to improve communication and teamwork and to increase vaginal delivery rates at hospital in the United States

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of a pilot project to improve communication and teamwork and to increase vaginal delivery rates at hospital in the United States. TeamBirth is a rigorously designed care process to improve care and SDM across the full care team, which includes the patient, their support person(s), nurse and physician or midwife, by ensuring reliability for best practices in communication and teamwork during labor and delivery. TeamBirth aims to operationalize best practices in communication and clinical care from the major professional organizations in obstetrics, including the American College of Obstetricians & Gynecologists (ACOG), Society for Maternal-Fetal Medicine (SMFM), American College of Nurse-Midwives (ACNM), and Association of Women's Health, Obstetric, and Neonatal Nurses (AWHONN), to ensure these practices are occurring consistently throughout labor. Key TeamBirth practices include:

1. Promoting the roles of the laboring patient, nurse, and delivering provider as members of the care team with equally valuable input for SDM,
2. Eliciting the patient's preferences, symptoms, and subjective experiences and integrating them with clinical data to inform patient care plans,
3. Distinguishing statuses and care plans for the mother, fetus, and labor progress, and
4. Setting shared expectations for the next planned evaluation.

ELIGIBILITY:
Clinician Participant Inclusion Criteria:

* All clinicians who have practice privileges at a study site

Clinician Participant Exclusion Criteria:

* None

Implementation Team Participant Inclusion Criteria:

* Champions, super-users and others who have been involved in the implementation of "Team Birth Project" at a study site

Implementation Team Participant Exclusion Criteria:

* None

Patient Participant Inclusion Criteria:

* 18 years or older
* Live birth. Includes: spontaneous or induction of labor; Vaginally, with an instruments (forceps / vacuum), or unscheduled cesarean delivery
* Patient at a study site piloting "Team Birth Project"

Patient Participant Exclusion Criteria:

* Under 18 years old
* Scheduled cesarean delivery
* Experienced intrapartum, stillbirth, or neonatal death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5217 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Weiseth, DNP, RN, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (4):
- United States (4):
  - South Shore Hospital, Weymouth, Massachusetts
  - Saint Francis Hospital, Tulsa, Oklahoma
  - Overlake Medical Center, Bellevue, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinicians: All nurses, midwives, and obstetricians in the participating units were invited to complete surveys using online links/QR codes; Patients: All patients >= 18 years (except Saint Francis where patients >= 15 years were included) who did not have a fetal demise or scheduled cesarean delivery were eligible during their postpartum stay
Pre-assignment Details: N/A for single group assignment
Period: Overall Study
Arm/Group | Implemented Health Facility
Started | 5217
Patients | 3924
Clinicians | 1293
Completed | 5217
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who consented to participate in patient or clinician surveys for the Team Birth Project; individual demographics were not captured for clinicians so all clinician participants are classified as "Unknown or Not Reported"
Arm/Group | Implemented Health Facility
Number analyzed (Participants) | 5217
Age, Customized [Count of Participants; unit: Participants]
  Age: Under 20 years old | 79
  Age: 20 - 24 years old | 443
  Age: 25 - 29 years old | 1105
  Age: 30 - 34 years old | 1439
  Age: 35 - 39 years old | 707
  Age: 40 years old or older | 107
  Age: Unknown or Not Reported | 1337
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 3924
  Gender: Male | 0
  Gender: Unknown or Not Reported | 1293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 325
  Not Hispanic or Latino | 3599
  Unknown or Not Reported | 1293
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 568
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 167
  White | 2563
  More than one race | 539
  Unknown or Not Reported | 1370
Region of Enrollment [Number; unit: participants]
  United States | 5217

OUTCOME MEASURES:

1. Primary Outcome: Percent of Clinicians Recommending TeamBirth Project
Description: At the project midline, percent of clinicians (physicians, midwives, and nurses) who would definitely or probably recommend the Team Birth project tools for use in other labor and delivery units.
Time Frame: The window begins on the 180th day to the 270th day from the start date at each site (180 days to 270 days). If clinicians complete more than one survey in the window, we will use the first one.
Population: Eligible clinicians (physicians, midwives, and nurses) who responded to a survey during the outcome measure time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Implemented Health Facility
Number analyzed (Participants) | 375
Participants
  Definitely | 254
  Probably | 83
  Maybe | 25
  Probably Not | 13
  Definitely Not | 0

2. Primary Outcome: Percent of Patients With the Role They Wanted in Decision-Making
Description: At the project midline, percent of patients who definitely or somewhat had the role they wanted in making decisions about their labor, among patients who wanted to make collaborative decisions with clinicians.
Time Frame: The window begins on the 180th day to the 270th day from the start date at each site (180 days to 270 days). Patients were only offered the survey once within the window.
Population: Eligible patients who responded to a survey and wanted to make collaborative decisions with clinicians during the outcome measure time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Implemented Health Facility
Number analyzed (Participants) | 805
Participants
  Yes, definitely | 726
  Yes, somewhat | 68
  No | 5
  Don't know / no opinion | 4
  Prefer not to answer | 2

ADVERSE EVENTS:
Time Frame: Up to 18 months at the facility level
Description: Clinician, maternal (at time of survey), and neonate (at time of survey) participants were not monitored/assessed for deaths or AEs. As surveys for maternal participants were anonymous, deaths and AEs could not be ruled out for either maternal or neonate participants. Therefore, Severe Maternal Morbidity, Severe Unexpected Newborn Complications, and Other Adverse Events were monitored/assessed for the general maternal and neonate populations and are reported at the facility level.
Groups:
- General Maternal Population (Facility Level): Serious AEs and Other AEs were collected at the facility level for all patients admitted (inclusive of those enrolled and not enrolled in the study). As surveys were anonymous, data from the General Maternal Population are reported as it could not be ruled out that enrolled maternal participants were not affected by severe maternal morbidity as a Serious AE and/or postpartum hemorrhage and maternal blood transfusion as an Other AE. Severe maternal morbidity was defined as the composite maternal outcomes measure developed by the Centers for Disease Control and Prevention, which includes "unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health".
- General Neonate Population (Facility Level): Serious AEs and Other AEs were collected at the facility level for all neonates of admitted patients (inclusive of those enrolled and not enrolled in the study). As surveys were anonymous, data for the General Neonate Population is reported as it could not be ruled out that neonates of enrolled maternal patient participants were not affected by severe or overall unexpected newborn complications as a Serious AE or Other AE, respectively. Unexpected newborn complications was defined as the composite neonatal outcomes measure developed by the California Maternal Quality Care Collaborative and adopted by The Joint Commission, which includes "unexpected newborn complications among full term newborns with no preexisting conditions".
Arm/Group | General Maternal Population (Facility Level) | General Neonate Population (Facility Level)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 328/14286 | 260/11063
Other Adverse Events (participants affected / at risk) | 662/7716 | 50/3737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | General Maternal Population (Facility Level) (N=14286) | General Neonate Population (Facility Level) (N=11063)
Severe Maternal Morbidity (Pregnancy, puerperium and perinatal conditions) | 328 (328) | 0/0 (0) — Assessed only in general maternal population. Data were available from South Shore Hospital, Saint Francis Hospital, and Overlake Medical Center.
Severe Unexpected Newborn Complication Rate (General disorders) | 0/0 (0) | 260 (260) — Assessed only in general neonate population. Data were available from South Shore Hospital,Saint Francis Hospital, and Evergreen Health Medical Center.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | General Maternal Population (Facility Level) (N=7716) | General Neonate Population (Facility Level) (N=3737)
Post Partpartum Hemorrhage (Pregnancy, puerperium and perinatal conditions) | 569 (569) | 0/0 (0) — Assessed only in general maternal population. Data were available from Evergreen Health Medical Center.
Maternal Blood Transfusion (Pregnancy, puerperium and perinatal conditions) | 93 (93) | 0/0 (0) — Assessed only in general maternal population. Data were available from Evergreen Health Medical Center.
Overall Unexpected Newborn Complication Rate (General disorders) | 0/0 (0) | 50 (50) — Assessed only in general neonate population. Data were available from Overlake Medical Center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03529214/Prot_SAP_000.pdf